CLINICAL TRIAL: NCT07187180
Title: Evaluating the Clinical Efficacy of Thulio vs. Holmium Laser Enucleation of the Prostate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Smita De (Other)
Responsible Party: Sponsor-Investigator, Smita De, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-209
Record Dates: First submitted 2025-06-16; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: BPH With Symptomatic Lower Urinary Tract Symptoms; BPH With Urinary Obstruction
Keywords: BPH; Enlarged prostate; Thulio laser; Prostate enucleation; male urinary retention
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control - Holmium (Active Comparator): Holmium laser enucleation
  Interventions: Device: holmium laser
- Experimental - Thulio (Experimental): Thulio laser enucleation
  Interventions: Device: pulsed thulium laser

INTERVENTIONS:
Device: holmium laser — Prostate enucleation will holmium laser (control)
  Arms: Control - Holmium
Device: pulsed thulium laser — experimental group - pulsed thulium laser prostate enucleation
  Arms: Experimental - Thulio

SUMMARY:
Many consider laser enucleation of the prostate the new 'gold standard' for the surgical treatment of benign prostatic hyperplasia (BPH) due to its excellent outcomes, high success rates, and long-term efficacy. Holmium laser enucleation of the prostate (HoLEP) was the earliest form of prostate enucleation and is recommended by the American Urological Association (AUA), along with thulium laser enucleation of the prostate (ThuLEP), as size-independent techniques for the management of BPH with fewer complications than transurethral resection of the prostate (TURP). Further development of laser technology has additionally led to enucleation using pulsed-modulated (e.g. "Virtual Basket™" mode or MOSES™ mode) holmium lasers as well as the thulium fiber laser.

DETAILED DESCRIPTION:
Study Design This is a prospective randomized study to evaluate the differences in outcomes comparing the existing laser to a new laser among patients undergoing HoLEP. Patients will be evaluated prior to the procedure and at one follow-up time point. Patients will be randomized in equal numbers to each group. The primary outcome will be non-inferiority in hemostasis timing. Several secondary outcomes will be evaluated including enucleation time, active laser time, morcellation time, prostate volume, change in hemoglobin, applied total laser energy, enucleation efficacy (g/min), IPSS (International Prostate Symptom Score), QoL (Quality of Life), uroflowmetry, PVR (post-void residual), duration of catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Patients must be males with a prostate, at least 18 years of age
* No prior prostate surgery

Exclusion Criteria:

* Unable/refuse to provide informed consent
* Prior prostate surgery
* Bladder stones that requiring lasering (small stone that can be removed whole is ok)
* Unable to hold anticoagulants or antiplatelets per standard protocols for surgery and up to 1 week postop.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Hemostasis time | During surgery
  time required to get adequate hemostasis intraoperatively

SECONDARY OUTCOMES:
Blood Loss | During surgery
  Estimated blood loss (mL)
Blood Loss | During surgery
  Change in hemoglobin (delta g/dL)
Operative parameters | During surgery
  Enucleation time (minutes)
Operative parameters | During surgery
  morcellation time (minutes)
Operative parameters | During surgery
  enucleation efficiency (mL prostate)
Laser parameters | During surgery
  Laser time (minutes)
Laser parameters | During surgery
  laser energy (joules)
Laser parameters | During surgery
  Fiber burn-back (cm)
Subjective laser performance | During surgery
  Surgeon estimation of collateral tissue injury and overall performance (scale 1 minimum 10 maximum)
Perioperative outcomes | 0-5 days after surgey
  volume of tissue removed (mL)
Perioperative outcomes | 0-5 days after surgery
  catheter time (hours)
Perioperative outcomes | 0-5 days after surgery
  length of stay (hours)
Perioperative outcomes | 30 days post op
  operative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Main, Cleveland, Ohio, United States

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-08-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT07187180/SAP_000.pdf